CLINICAL TRIAL: NCT06336915
Title: Physician-Nurse Dyad Rounding: A Collaborative Approach to Improve Unit-Level Metrics
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 121.NUR.2022.D
Record Dates: First submitted 2023-03-30; First posted 2024-03-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Wellness, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Physician-Nurse Dyad Rounding — Collaborative Approach to Improve Unit-Level Metrics

SUMMARY:
The project will be implemented on one unit at a time until the co-rounding process has been implemented on each Medical-Surgical unit. This study will involve the geo-localized hospitalist on the designated unit and the nursing staff involved in clinical patient care

DETAILED DESCRIPTION:
Patient experience top box scores as well as doctor and nurse domains will be evaluated retrospectively prior to project implementation and this evaluation will continue to be evaluated six months after IRB approval and project initiation. Baseline patient experience scores are routinely captured as a part of routine data collection practices via Press Ganey survey administration.

LOS and discharge times are also routinely collected as a part of routine data collection practices. LOS and average discharge times will be reviewed on an ongoing basis after project implementation to monitor for improvements.

ELIGIBILITY:
Inclusion Criteria:

* Patient Experience, LOS, and Discharge Times: Private hospitalist patients at MDMC
* LOS: Patients with a LOS ≤20 days

Exclusion Criteria:

* Patient Experience: Patients other than private hospitalist patients excluded from this measure.
* LOS: Patients with LOS >20 days are considered an outlier and will be excluded from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Private hospitalist patients at MDMC
  Patients with a LOS ≤20 days
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Difference in percentage of discharged patients before 1400 (Mon-Fri) after project implementation compared to before implementation | "up to 100 weeks"
  Difference in percentage of discharged patients before 1400 (Mon-Fri) after project implementation compared to before implementation

SECONDARY OUTCOMES:
Difference in Top Box Patient Satisfaction Scores and Doctor Domain | "up to 100 weeks"
  Difference in top box patient satisfaction scores and doctor domain for private hospitalist patients after project implementation compared to before implementation
Difference in LOS of private hospitalist patients after project implementation compared to before implementation | "up to 100 weeks"
  Difference in LOS of private hospitalist patients after project implementation compared to before implementation
Difference in collaboration and build positive relationships scores after project implementation compared to before implementation | "up to 100 weeks"
  Difference in collaboration and build positive relationships scores after project implementation compared to before implementation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Research Institute at Methodist Health System, Dallas, Texas
  - Methodist Dallas Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All study-related documents will be retained by the CRI until at least three years after study completion or according to local laws, whichever is longer
Access Criteria: Records will also be accessible to MHS staff upon request unless constituting a violation of patient confidentiality

REFERENCES:
- [Background] Pritts KE, Hiller LG. Implementation of Physician and Nurse Patient Rounding on a 42-Bed Medical Unit. Medsurg Nurs. 2014 Nov-Dec;23(6):408-13. PMID 26281644
- [Background] Shortell, S. (1989). ICU Nurse Questionnaire. Excerpted from The Organization and Management of Intensive Care Units. Copyright 1989, Shortell and Rousseau.
- [Background] Rigel, N., Delp, S., Ward, C. (2018). Effects of Nurse-Physician Collaborative Rounding, MEDSURG Nursing, 27(3) 149-152.
- [Background] Sturdivant, T., Herrin, K., Reynolds, M., Mestas, L. (2020). Improving Patient Satisfaction through a Nurse Leader-Physician Bedside Rounding Protocol: A Pilot Project, Nursing Econonmic$, 38(3).